CLINICAL TRIAL: NCT00984425
Title: Phase I and Pharmacokinetics Study of Lapatinib in Combination With Sorafenib in Patients With Advanced Refractory Solid Tumors
Brief Title: The Treatment of Lapatinib in Combination With Sorafenib in Patients With Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2008-005
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Lapatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lapatinib and Sorafenib 1° level of dose (Experimental): Lapatinib 750 mg/die + Sorafenib 200 mg bid
  Interventions: Drug: Lapatinib and Sorafenib
- Lapatinib and Sorafenib 2° level of dose (Experimental): 2° level (II cohort): Lapatinib 1000 mg/die + Sorafenib 200 mg bid
  Interventions: Drug: Lapatinib and Sorafenib
- Lapatinib and Sorafenib 3° level of dose (Experimental): 3° level (III cohort): Lapatinib 1000 mg/die + Sorafenib 400 mg bid
  Interventions: Drug: Lapatinib and Sorafenib
- Lapatinib and Sorafenib 4° level of dose (Experimental): 4° level (IV cohort): Lapatinib 1250 mg/die + Sorafenib 400 mg bid
  Interventions: Drug: Lapatinib and Sorafenib

INTERVENTIONS:
Drug: Lapatinib and Sorafenib — Comparison of different dosages of two drug
  Other Names: Tykerb and Nexavar

SUMMARY:
Over the last decade, improvements in the investigators' understanding of the molecular basis of cancer have led to the clinical development of protein kinase inhibitors, which target pivotal molecules involved in intracellular signaling pathways implicated in tumorigenesis and tumor progression. Lapatinib is an oral selective and reversible inhibitor of the tyrosine kinase domain of epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor type 2 (HER-2), which are both frequently altered in human malignant tumors. Sorafenib is an oral multi-kinase inhibitor with a dual-action that prevents tumor cell proliferation and angiogenesis. The investigators suggest that through a complete blockade of ErbB signaling network it may be possible to ''sensitize'' tumor cells to antiangiogenic therapy, by lowering the tumor cell survival threshold, while through inhibition of vascular endothelial growth factor (VEGF) pathway to circumvent the problem of acquired resistance to EGFR inhibitors. Based on this theoretical rationale we decide to test the combination of Lapatinib and Sorafenib. This phase I trial will be undertaken to assess the maximum dose tolerated (MTD), safety/tolerability, pharmacokinetics and antitumor efficacy of this combination in patients with advanced, recurrent or metastatic solid cancers refractory to available standard treatment.

DETAILED DESCRIPTION:
This is a dual-agent, prospective, open-label, multi-centric, phase I trial of combination of Lapatinib and Sorafenib in patients with locally advanced, recurrent or metastatic solid tumors. This trial will be conducted to determine the maximum tolerated dose (MTD), safety/tolerability, pharmacokinetics, and antitumor activity of these two agents given together on a continuous schedule, in patients with advanced solid tumors.

Our ambition is to recommend a safe dose regimen of the combination for subsequent larger phase II studies, coinciding with the maximum tolerated dose (MTD).

The maximum tolerated dose (MTD), will be defined as the highest dosage cohort at which no more than one of six patients will be experienced a DLT in the first treatment cycle.

Eligible patients will be enrolled and treated according to the schema, using a 3+3 design (Fibonacci method modified);

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced, recurrent or metastatic histologically confirmed malignancy refractory to available standard treatment

Exclusion Criteria:

* Prior treatment with Lapatinib, Sorafenib or any agents targeting EGFR (other than trastuzumab), Raf, VEGF, or VEGFR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities (DLTs)and the maximum tolerated dose (MTD) of the combination of Lapatinib and Sorafenib. | 0ne year

SECONDARY OUTCOMES:
To determine the safety profile of escalating doses of Lapatinib in combination with escalating doses of Sorafenib and and to compare the pharmacokinetics of Lapatinib alone and in combination with Sorafenib | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Result] Simonelli M, Zucali PA, Lorenzi E, Rubino L, De Vincenzo F, De Sanctis R, Perrino M, Mancini L, Di Tommaso L, Rimassa L, Masci G, Zuradelli M, Suter MB, Bertossi M, Fattuzzo G, Giordano L, Roncalli MG, Santoro A. Phase I pharmacokinetic and pharmacodynamic study of lapatinib in combination with sorafenib in patients with advanced refractory solid tumors. Eur J Cancer. 2013 Mar;49(5):989-98. doi: 10.1016/j.ejca.2012.10.016. Epub 2012 Nov 9. PMID 23146956